CLINICAL TRIAL: NCT00542074
Title: Bacterial Vaginosis; A Randomized Trial to Reduce Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-9276-001; R03TW005820 (NIH); HD 40540-04; P30AI027757 (NIH)
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial vaginosis; recurrence; male factor
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence | interventions — Ethanol; hydroxide ion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: hygienic information plus 62% ethyl alcohol in emollient gel
- 2 (Active Comparator)
  Interventions: Other: hygienic information

INTERVENTIONS:
Other: hygienic information plus 62% ethyl alcohol in emollient gel — The male partner in each couple was asked to apply Purell® to his penis at least daily, and immediately prior to and following intercourse. Couples received a brochure with information on control of STI and good hygienic practices. Brochures for intervention and control arms were similar except the intervention arm brochure provided information on how to use the study product (Purell®).
  Other Names: Purell® (GOJO Healthcare Inc., Akron, OH)
  Arms: 1
Other: hygienic information — Couples received a brochure with information on control of STI and good hygienic practices.
  Arms: 2

SUMMARY:
Randomized controlled trial (RCT) to evaluate the effectiveness of applying Purell® (62% ethyl alcohol in emollient gel) to the penis of male partners of women diagnosed with BV for preventing BV recurrence after treatment.

ELIGIBILITY:
Inclusion criteria:

* Vaginal symptoms
* Nugent score > 6 for vaginal fluid gram stain
* Woman and her male partner both interested in study participation
* Woman able to return for follow-up visits
* Woman able to provide detailed contact information for tracing

Exclusion Criteria:

* Either male or female partner not recruited within 24 hours of the other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2003-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
bacterial vaginosis by Nugent's score | up to 2 months following treatment

SECONDARY OUTCOMES:
presence of lactobacillus by culture | 2 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: King K. Holmes, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Nairobi City Council STI referral clinic (Special Treatment Clinic), Nairobi, Kenya